CLINICAL TRIAL: NCT01524497
Title: A Clinical Study on Efficacy And Safety of Trazodone Hydrochloride Prolonged-Release Tablets for Treatment of Depression A Multicenter, Randomized, Double-Blind, Parallel Controlled Study
Brief Title: A Clinical Study of Trazodone Hydrochloride Prolonged-Release Tablets for Treatment of Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trazodone_1
Record Dates: First submitted 2012-01-13; First posted 2012-02-02 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: losing interest and feelings of guilt; poor concentration; loss of appetite; suicide
MeSH Terms: conditions — Depression; Anorexia; Suicide | interventions — Trazodone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trazodone (Active Comparator)
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trazodone — 75mg tablet/150 mg tablet
  Arms: Trazodone
Drug: Placebo — Reference drug: trazodone hydrochloride prolonged-release tablet placebo (corresponding dummy drug of 75mg, 150mg active drug)
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the efficacy and safety of trazodone hydrochloride prolonged-release tablets for treatment of depression in Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65, males and females, outpatients or inpatients;
2. Single episode or recurrent depression according to DSM-IV (Version 4) criteria;
3. Scores > 18 on 17-item HAM-D at screening and baseline visits with a decrease not exceeding 20% between the two visits;
4. Symptoms of depression for at least 1 month;
5. Patients or their dependents/guardians providing signed informed consent forms.

Exclusion Criteria:

1. Serious suicide attempts (≥ 3 on item 3 'Suicide' of HAMD);
2. Depressive episode, with psychotic symptoms;
3. Refractory depression;
4. Depressive episode secondary to other mental or physical disorders;
5. Bipolar disorder;
6. Significant reduction in body weight and malnutrition induced by major depression;
7. Serious or unstable heart, hepatic, renal, endocrine and hematologic disease or malignant tumors;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 score | six weeks
  17-item Hamilton Depression Rating scale were evaluated at the basemline and six weeks after treatment, the changes were recorded and used as primary outcome measurement.

SECONDARY OUTCOMES:
Changes in HAMA-14 score | Six weeks
  Change from baseline in HAMA-14 score at Visit 6/final visit
CGI-Severity of illness and CGI-Global improvement | Six weeks
  CGI-Severity of illness and CGI-Global improvement at Visit 6/final visit
Changes in evaluation of sleep quality and sexual dysfunction | Six weeks
  change from baseline in evaluation of sleep quality and sexual dysfunction at Visit 6/final visit
Rate changes of responders/patients | Six weeks
  rate of responders, defined as patients with a 50% improvement from baseline in the HAMD score at Visit6/final visit;or rate of patients with remission, defined as patients with HAMD score ≤7 at Visit 6/final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin LI, Ph.D., Study Director — Lee's Pharmaceutical company
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China